CLINICAL TRIAL: NCT03987984
Title: Reliability and Validity of the Turkish Version of the Sensory Eating Problems Scale (VERSION)
Brief Title: Reliability and Validity of the Turkish Version of the Sensory Eating Problems Scale
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Muserrefe Nur Keles, PhD, PT, Research Assistant, Gazi University
Other Study IDs: 19882019
Record Dates: First submitted 2019-06-14; First posted 2019-06-17 (Actual); Last update posted 2021-10-15 (Actual); Status verified 2021-10

CONDITIONS: Feeding and Eating Disorders
Keywords: Sensory Feeding Problems
MeSH Terms: conditions — Feeding and Eating Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study was to adapt to the Sensory Eating Problems Scale to Turkish. Within the scope of the study, firstly the Turkish version of the scale will be developed and then its reliability and validity will be examined.

DETAILED DESCRIPTION:
The etiology of childhood feeding problems is often complex and likely due to multiple factors, such as biological issues, oral motor deficits, and environmental contingencies. Sensory processing, or the ability to receive, integrate, and process sensory input, such as visual, olfactory, or gustatory information, has also been speculated to influence eating. A growing literature has examined the association between sensory processing and eating behavior in several populations of children.

While child feeding problems have been found to be associated with withsensory processing problems, clinicians could benefit from more specifics about the types of oral sensory problems most associated with feeding problems. For example, the Oral Sensory Processing subscale of the Sensory Profile includes a collection of sensory problems associated with feeding difficulties such as gagging easily to food or utensils in the mouth, rejecting certain food tastes or smells, accepting limited food textures, biting the tongue or lips , but without documentation that identifies the separate dimensions of oral sensitivity problems relevant to children's feeding problems. Further, along theOral Sensory Processing Subscale of the SP, a particular oral sensory problems, such as sensitivity to texture, may be measured by only one or two items.

Sensory Eating Problems Scale is a newly developed scale and can measure specific oral sensory problems in children. SEPS can also provide a more detailed assessment of sensory eating behavior than provided in previous studies by developing the Sensory Eating Problems Scale (SEPS) to identify specific dimensions of oral sensitivity children show during feeding. However; there is no short, easy to use and easy to understand sensory eating problems scale with the Turkish version.

ELIGIBILITY:
Inclusion Criteria:

* The children had been referred to the clinics for eating problems that included failure to gain weight, dependence on tube feeding or oral supplements, difficulties with texture or learning to chew, limited diet variety, and mealtime behavior problems.

Exclusion Criteria:

-

Ages: 2 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children with 2-6 years and have eating problems that included failure to gain weight, dependence on tube feeding or oral supplements, difficulties with texture or learning to chew, limited diet variety, and mealtime behavior problems.
Sampling Method: Non-Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2019-06-14 (Actual); Primary Completion 2020-08-05 (Actual); Study Completion 2021-12-15 (Estimated)

PRIMARY OUTCOMES:
Sensory Eating Problems Scale | 2 weeks
  The 22-item scale developed in the present study offers clinicians and researchers a new measure to examine more specific sensory eating problems than other sensory profiles.

SECONDARY OUTCOMES:
Behavioral Pediatrics Feeding Assessment Scale | 2 weeks
  The scale is a widely used parent-report measure of meal time and feeding behavior. It consists of 35 items; the first 25 of which focus on child behavior and the last 10 of which provide an index of parental feelings about, and strategies for, addressing mealtime and feeding problems.
Caregiver reported Feeding/Swallowing Impact Survey | 2 weeks
  The survey was designed to evaluate caregivers' various responses to questions about quality of life related to activities of daily living, feeding, and generalized worry with 6 items in each category.

CONTACTS AND LOCATIONS:
Overall Officials: Müşerrefe N Keleş, PhD, Principal Investigator — Gazi University
Locations (1):
- Gazi University, Faculty of Health and Sciences, Department of Physiotherapy and Rehabilitation, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No